CLINICAL TRIAL: NCT05866081
Title: Stent Omission After Ureteroscopy and Lithotripsy in the Michigan Urological Surgery Improvement Collaborative (SOUL MUSIC)
Brief Title: Stent Omission After Ureteroscopy and Lithotripsy in the Michigan Urological Surgery Improvement Collaborative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Michigan Urological Surgery Improvement Collaborative (MUSIC) (Other)
Responsible Party: Principal Investigator, Khurshid Ghani, Professor of Urology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00234740; CER-2021C2-22856 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stone, Kidney; Stone Ureter
Keywords: Unilateral ureteroscopy and lithotripsy; Ureteral stent; Pain assessment; Quality of life
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants that consent for the randomization cohort (264 anticipated) will be randomized using an online computer-based system to either stent omission or stent placement in a 1:1 ratio following secondary eligibility criteria. Blocked, stratified randomization based upon surgeon classified stone location (renal only versus ureteral with or without renal), with random block sizes will be used to ensure group balance.
  Observational study participants (528 anticipated) will not be randomized.
Who Masked: Care Provider
Masking Description: Surgeons will remain blinded to this allocation until the surgeon has confirmed secondary eligibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Randomized cohort- No stent placement (Other): Participants that are eligible and consent for the randomization cohort of the trial will not have a stent placed.
  If participants are found to be ineligible (see below) at the end of ureteroscopy the participants will not be randomized and taken off the study.
  In randomization cohort, second stage eligibility criteria: ureteral perforation, unanticipated anatomic abnormality, greater than expected bleeding, ureteral dilation greater than 12 French, ureteral access sheath utilized, failed ureteroscopy, no or incomplete lithotripsy performed, unable to complete case due to medical or anesthetic event.
  Interventions: Other: No stent placement; Other: Surveys
- Randomized cohort- Stent placement (Experimental): Participants that are eligible and consent for the randomization cohort trial will have a stent placed.
  If participants are found to be ineligible (see below) at the end of ureteroscopy the participants will not be randomized and taken off the study.
  In randomization cohort, second stage eligibility criteria: ureteral perforation, unanticipated anatomic abnormality, greater than expected bleeding, ureteral dilation greater than 12 French, ureteral access sheath utilized, failed ureteroscopy, no or incomplete lithotripsy performed, unable to complete case due to medical or anesthetic event.
  Interventions: Device: Standard of care stent placement; Other: Surveys
- Observational participants - not randomized (Other): Patients that do not consent to the randomization trial that elect to be on the observational cohort. Stent placement in the observational cohort will be decided by the surgeon intraoperatively, as per routine clinical practice.
  Interventions: Other: Surveys

INTERVENTIONS:
Device: Standard of care stent placement — Participants will have a stent placed per randomization assigned if there are no complications (per protocol) during ureteroscopy that excludes the participant.
  Arms: Randomized cohort- Stent placement
Other: No stent placement — Participants not have a stent placed per randomization assigned if there are no complications (per protocol) during ureteroscopy that excludes the participant.
  Arms: Randomized cohort- No stent placement
Other: Surveys — All participants in the trial cohort and observational arms will be asked to complete survey instruments (evaluating their pain, quality of life, and experiences following ureteroscopy, as well as surveys evaluating their opinions and preferences around ureteral stenting, etc.).
  Participants will also have routine clinical data (preoperative, perioperative, and postoperative) to be collected and analyzed for research purposes.

SUMMARY:
This is a multicenter prospective trial with randomized and observational cohorts assessing patient-reported outcomes and unplanned healthcare utilization following ureteroscopic treatment of renal and ureteral stones, with placement versus omission of a ureteral stent.

Eligible participants in the randomization trial will be randomized to ureteroscopy with stent placement or stent omission.

Eligible participants that consent to the observational only cohort will complete surveys and the treating physicians will decide the treatment options for the participants.

The study team hypothesizes that:

* Pain interference change from pre-surgery to Day 7-10 will differ between the two treatment arms. This hypothesis will be evaluated separately in the randomized and observational cohorts.
* Unplanned healthcare utilization in the treatment arms will have different unplanned healthcare utilization ranks leading to a win proportion significantly higher or lower than 0.5 in the stent omission arm compared to the stent placement arm. This hypothesis will be evaluated separately in the randomized and observational cohorts.

DETAILED DESCRIPTION:
The coordinating center for this study is the Michigan Urological Surgery Improvement Collaborative (MUSIC), which is a physician-led Quality Improvement (QI) collaborative comprised of 44 urology practices and 260 urologists across the State of Michigan.

As sites are activated the registration will be updated.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing unilateral ureteroscopy and lithotripsy for stone disease (participants may have contralateral stones, as long as these are asymptomatic and not being treated concurrently)
* Largest stone less or equal to 10 millimeter in size as measured on abdominal x-ray, ultrasound, or computed tomography scan
* Access to means of communication with the study team (email, text messaging, and/or telephone)
* Adequate independent cognitive function and English language proficiency to complete study surveys
* Written informed consent

Exclusion Criteria:

* Planned bilateral ureteroscopy
* Indwelling ureteral stent or percutaneous nephrostomy tube preoperatively in either kidney
* Anatomic abnormalities of the ipsilateral upper urinary tract (for example, horseshoe kidney, crossed fused ectopia, pelvic kidney, urinary diversion)
* Anatomic or functional solitary kidney
* Planned secondary or staged ureteroscopy
* Planned use of ureteral access sheath
* Pregnancy
* Patients who use opiate medication daily for greater than 3 months to manage a painful condition

Second Stage Exclusion Criteria:

* ureteral perforation
* unanticipated anatomic abnormality
* greater than expected bleeding
* ureteral dilation greater than 12 French
* ureteral access sheath utilized
* failed ureteroscopy
* no or incomplete lithotripsy performed
* unable to complete case due to medical or anesthetic event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS®) Pain Interference (Short Form 6b) change at Postoperative Day 7-10 compared to preoperative | Preoperative, Day 7-10
  This survey has 6 questions that participants select from 1(not at all) to 5 (very much) for questions 1-5 related to pain interference. For question 6 participants select from 1 (Never) to 5 (Always). There are total of 6-30 points where the higher the score the more pain interference.
Number of Participants with Wins from the Hierarchical Unplanned stone treatment related healthcare utilization Composite Rank Score | within 30 days after ureteroscopy
  Compare within each cohort each No Stent Placement patient head-to-head against each Stent Placement patient using a hierarchical composite comprised of:
  * Intensive care unit (ICU) care during hospitalization
  * Unplanned hospitalization
  * Unplanned additional procedure related to ureteroscopy: operating room or interventional radiology procedure
  * Emergency department visit
  * Unplanned clinic visit and/or diagnostic testing (blood, urine testing and/or imaging)
  * Number of ambulatory patient-provider interactions: phone calls / Electronic Medical Record (EMR) messages

SECONDARY OUTCOMES:
Number of Participants with Intensive Care Unit care during unplanned hospital admission within postoperative day 30 | within 30 days after ureteroscopy
Number of Participants with Unplanned hospital admission within postoperative day 30 | within 30 days after ureteroscopy
Number of Participants with Unplanned additional procedure related to ureteroscopy within postoperative day 30 | within 30 days after ureteroscopy
Number of Participants with Unplanned ambulatory urology office visit and/or diagnostic testing (urine testing and/or imaging) within postoperative day 30 | within 30 days after ureteroscopy
Unplanned ambulatory urology office visit and/or diagnostic testing (urine testing and/or imaging) within postoperative day 30 | within 30 days after ureteroscopy
Number of ambulatory patient-provider interactions: phone calls / EMR messages within postoperative day 30 | within 30 days after ureteroscopy
PROMIS® Pain Interference (Short Form 6b) change at postoperative 4-6 weeks compared to preoperative | preoperative, 4-6 weeks
  This survey has 6 questions that participants select from 1(not at all) to 5 (very much) for questions 1-5 related to pain interference. For question 6 participants select from 1 (Never) to 5 (Always). There are total of 6-30 points where the higher the score the more pain intensity.
PROMIS® Pain Intensity (Short Form 3a) change at postoperative day 7-10 preoperative | preoperative, postoperative day 7-10
  This is a 3-question survey that participants select from 1 (had no pain) to 5 (very severe) for the first 2 questions. For the third question participants select how level of pain is now 1 (no pain) to 5 (very severe). There are total of 3-15 points where the higher the score the more pain intensity.
PROMIS® Pain Intensity (Short Form 3a) change at postoperative 4-6 weeks compared to preoperative | preoperative, postoperative 4-6 weeks
  This is a 3-question survey that participants select from 1 (had no pain) to 5 (very severe) for the first 2 questions. For the third question participants select how level of pain is now 1 (no pain) to 5 (very severe). There are total of 3-15 points where the higher the score the more pain interference.
National Institutes of Health (NIH) Lower Urinary Tract Dysfunction Research Network (LURN) Symptom Index-10 urinary symptom scores change at postoperative day 7-10 compared to preoperative | preoperative, postoperative day 7-10
  The is 10-Item index that assesses participants urinary symptoms. For questions 1-8 Participants select from 0 (never)-4 every time. For questions 9 and 10 participants select from 0 (none) -3 (more than 3 times). There are total of 0-38 points where the higher the score the more pain symptoms.
National Institutes of Health (NIH) Lower Urinary Tract Dysfunction Research Network (LURN) Symptom Index-10 urinary symptom scores change at postoperative 4-6 weeks compared to preoperative | preoperative, postoperative 4-6 weeks
  The is 10-Item index that assesses participants urinary symptoms. For questions 1-8 Participants select from 0 (never)-4 every time. For questions 9 and 10 participants select from 0 (none) -3 (more than 3 times). There are total of 0-38 points where the higher the score the more pain intensity.
International Consultation on Incontinence - Satisfaction (ICIQ-S) treatment satisfaction scores at postoperative day 7-10 | Postoperative day 7-10
  Participants will complete this 14-question survey regarding satisfaction of treatment.
  The ICIQ-S assesses aspects of experience, expectations, and outcomes to evaluate satisfaction after urological surgery. A scoring system has been derived that consists of two parts: a score for the evaluation of satisfaction with 'surgical outcomes' (ICIQ-S outcome score, range 0-24); and the overall satisfaction with surgery item, scored 0-10. Higher scores indicate more satisfaction.
International Consultation on Incontinence - Satisfaction (ICIQ-S) treatment satisfaction scores at postoperative 4-6 weeks | Postoperative 4-6 weeks
  Participants will complete this 14-question survey regarding satisfaction of treatment.
  The ICIQ-S assesses aspects of experience, expectations, and outcomes to evaluate satisfaction after urological surgery. A scoring system has been derived that consists of two parts: a score for the evaluation of satisfaction with 'surgical outcomes' (ICIQ-S outcome score, range 0-24); and the overall satisfaction with surgery item, scored 0-10. Higher scores indicate more satisfaction.
Number of days taken off work by patients and caregivers during the first 7 days after ureteroscopy | First 7 days after ureteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid Ghani, MD, Principal Investigator — University of Michigan
Locations (16):
- United States (16):
  - University of Arizona, Tucson, Arizona
  - UF Health Shands Hospital, Gainesville, Florida
  - Indiana University Department of Urology, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan Health System, Brighton, Michigan
  - Cadillac Munson Hospital, Cadillac, Michigan
  - St. Joseph Health System Chelsea Hospital, Chelsea, Michigan
  - St. Joseph Mercy Health (Trinity), Chelsea, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Corewell Health Buttersworth Hospital, Grand Rapids, Michigan
  - E.W Sparrow Hospital, Lansing, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Michigan Institute of Urology Town Center Ambulatory Surgery Center, Troy, Michigan
  - Monte Fiore, Brooklyn, New York
  - Mount Sinai, New York, New York
  - UNC Hospital, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker REN, Daignault-Newton S, Shoemaker E, Sitek D, Thelus JM, Clark S, Martin-Schwarze A, Spino C, Carlozzi NE, Meurer WJ, Sales AE, Dauw CA, Ghani KR. Stent Omission after Ureteroscopy and Lithotripsy (SOUL) in the Michigan Urological Surgery Improvement Collaborative (MUSIC): study protocol for a pragmatic prospective combined randomized and observational clinical trial. Trials. 2024 Dec 4;25(1):811. doi: 10.1186/s13063-024-08587-8. PMID 39633425